CLINICAL TRIAL: NCT05764798
Title: Shugan Jieyu Capsule for Insomnia Patients With Depressive Symptoms: A Randomized Double Blind Controlled Study
Brief Title: Shugan Jieyu Capsule for Insomnia Patients With Depressive Symptoms
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2023-030
Record Dates: First submitted 2023-02-19; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Shugan Jieyu Capsule combined with zolpidem (Experimental): Zolpidem was given orally for basic treatment, with the treatment dose of 10mg/tablet per day, one tablet per time, once a day, before sleep, for 8 consecutive weeks. Shugan Jieyu Capsule was given orally, with a therapeutic dose of 0.36g/capsule, 2 capsules each time, twice a day, and once after breakfast and dinner.
  Interventions: Drug: Experimental group: Shugan Jieyu Capsule combined with zolpidem
- Control group: Placebo combined with zolpidem (Placebo Comparator): Zolpidem was given orally for basic treatment, with the treatment dose of 10mg/tablet per day, one tablet per time, once a day, before sleep, for 8 consecutive weeks. Placebo was given orally, with a therapeutic dose of 0.36g/capsule, 2 capsules each time, twice a day, and once after breakfast and dinner.
  Interventions: Drug: Control group: Placebo combined with zolpidem

INTERVENTIONS:
Drug: Experimental group: Shugan Jieyu Capsule combined with zolpidem — Shugan Jieyu capsule and zolpidem orally for 8 consecutive weeks
  Arms: Experimental group: Shugan Jieyu Capsule combined with zolpidem
Drug: Control group: Placebo combined with zolpidem — Placebo and zolpidem orally for 8 consecutive weeks
  Arms: Control group: Placebo combined with zolpidem

SUMMARY:
This study is a randomized, placebo-controlled, double-blind clinical study. 60 cases of insomnia patients with depressive symptoms are planned to be treated, and they are randomly assigned to the experimental group (Shugan Jieyu Capsule combined with zolpidem group) and the control group (placebo combined with zolpidem group) in equal proportion. Both groups are given zolpidem orally for basic treatment, with the treatment dose of 10mg per tablet per day, one tablet per time, once a day, before sleep, for 8 consecutive weeks. The test group was given Shugan Jieyu Capsule orally, with a therapeutic dose of 0.36g per capsule, 2 capsules each time, twice a day, and once after breakfast and dinner. The control group was given placebo orally, with a treatment dose of 0.36g per capsule, 2 capsules each time, twice a day, and once after breakfast and dinner. The therapeutic effect of Shugan Jieyu Capsule on insomnia patients with depressive symptoms was observed by analyzing the changes of ISI scores, subjective and objective sleep indicators (PSG, sleep diary), daytime cognitive function, autonomic nervous function and EEG after the intervention in the fourth and eighth weeks.

ELIGIBILITY:
Inclusion Criteria:

* Conform to DSM-5 diagnostic criteria for insomnia.
* Moderate or above depressive symptoms: patient health questionnaire depression scale (PHQ-9) ≥ 10 points.
* No drug treatment for insomnia and/or depression within one month before the start of this study.
* 18-60 female or male.
* Can understand and comply with the research protocol, and can sign a written informed consent.

Exclusion Criteria:

* Shift workers, perennial night shift workers, frequent cross time zone pilots (such as crew members of international flights).
* PSG examination revealed sleep apnea syndrome (Apnea Hypopnea Index, AHI) ≥ 15 times one hour) and/or periodic limb movement disorder (periodic Limb Movement Index, PLMI] ≥ 15 times one hour).
* Those who have serious heart disease (such as heart failure, acute myocardial infarction, arrhythmia, coronary heart disease), liver disease (such as hepatitis, cirrhosis, liver cancer, alcoholic liver), lung disease (such as asthma, acute pneumonia, tuberculosis, lung cancer), kidney disease (such as acute and chronic glomerulonephritis, nephrotic syndrome) and other systemic diseases (such as diabetes) that need treatment.
* Have previously diagnosed mental disorders.
* Comply with DSM-5 diagnostic criteria for depression
* Allergic constitution, known or suspected of hypericum perforatum, acanthopanax senticosus and zolpidem allergy history.
* The past used of zolpidem or Shugan Jieyu capsule was ineffective.
* Liver function test ALT, AST>2 times the upper limit of reference value, or Scr>the upper limit of reference value.
* The P450 3A4 inhibitors of liver metabolic cytochrome enzyme have been used within 14 days before randomization, including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, acezotocin, indinavir, nafinavir, linavir, fluvoxamine, and saquinavir.
* The P450 3A4 inducer of liver metabolic cytochrome enzyme has been used within 14 days before randomization, including but not limited to phenytoin, carbamazepine, barbiturates, rifampicin, St. John's wort, and glucocorticoids.
* Substance or alcohol dependence (except complete remission and caffeine or nicotine dependence) according to DSM-IV standard at the time of inclusion.
* The abuse of opioids, amphetamines, barbiturates, cocaine, cannabis or hallucinogens according to DSM-IV standards 4 weeks before enrollment.
* Medical conditions that affect the absorption, distribution, metabolism or excretion of the study drug.
* Participated in clinical research of other drugs 4 weeks before enrollment or longer before enrollment according to actual requirements.
* Pregnant or lactating women.
* Those who committed serious suicide or committed suicide planning.
* Other situations unsuitable for inclusion in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index scale | Baseline and four, eight weeks after treatment
  Changes in insomnia severity index scale

SECONDARY OUTCOMES:
Pittsburgh sleep quality index scale | Baseline and four, eight weeks after treatment
  Changes in pittsburgh sleep quality index scale
Patient health questionnaire | Baseline and four, eight weeks after treatment
  Changes in patient health questionnaire
Facade severity scale | Baseline and four, eight weeks after treatment
  Changes in facade severity scale
Epworth sleeping scale | Baseline and four, eight weeks after treatment
  Changes in epworth sleeping scale
Polysomnography | Baseline and four, eight weeks after treatment
  Changes in the time to fall asleep, times of waking up at midnight and times of waking up early
Sleep diary | Baseline and four, eight weeks after treatment
  Changes in the time to fall asleep, the total time to wake up in the middle of the night and the time to wake up early
Generalized anxiety disorder scale | Baseline and four, eight weeks after treatment
  Changes in generalized anxiety disorder scale
Beck scale for suicide ideation--Chinese Version scale | Baseline and four, eight weeks after treatment
  Changes in beck scale for suicide ideation--Chinese Version scale
Concise happiness and quality of life satisfaction questionnaire | Baseline and four, eight weeks after treatment
  Changes in concise happiness and quality of life satisfaction questionnaire
Event-related potential | Baseline and four, eight weeks after treatment
  Changes in P300 latency
Heart rate variability analysis | Baseline and four, eight weeks after treatment
  Changes in low frequency, high frequency, very low frequency, low frequency/high frequency
N-back paradigm task | Baseline and four, eight weeks after treatment
  Changes in reaction time and accuracy
Suicide stroop task | Baseline and four, eight weeks after treatment
  Changes in reaction time and accuracy
Go/no-go association task | Baseline and four, eight weeks after treatment
  Changes in reaction time and accuracy
Psychomotor vigilance task | Baseline and four, eight weeks after treatment
  Changes in reaction time

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zhang, MD & PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xin Q, Paudel D, Zhang J, Wei H, Cheng Y, Xu Y, Fang R, Jiang J, Wang Y, Zhang B. Efficacy and safety of Shugan Jieyu capsules in combination with zolpidem for insomnia disorder with depressive symptoms: a double-blind randomized controlled trial. BMC Complement Med Ther. 2025 Oct 17;25(1):383. doi: 10.1186/s12906-025-05142-z. PMID 41107798